CLINICAL TRIAL: NCT02973711
Title: A Phase I/II Study of Ruxolitinib in Combination With Nilotinib in Patients With Chronic Phase CML Who Have Achieved a Complete Hematologic Remission, Complete Cytogenetic Remission, and Major Molecular Remission, But Not a Complete Molecular Remission on a Tyrosine Kinase Inhibitor Alone.
Brief Title: A Study of Ruxolitinib in Combination With Nilotinib in Patients With Chronic Phase CML
Status: Withdrawn | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: lack of funding
Sponsor: University of Michigan Rogel Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UMCC 2015.103; HUM00122063 (Other: University of Michigan)
Record Dates: First submitted 2016-11-22; First posted 2016-11-25 (Estimated); Last update posted 2021-02-16 (Actual); Status verified 2021-02

CONDITIONS: Leukemia, Chronic Myeloid
MeSH Terms: conditions — Leukemia, Myelogenous, Chronic, BCR-ABL Positive | interventions — nilotinib; ruxolitinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Nilotinib + Ruxolitinib (Experimental): The first part of the trial will be Phase I and will enroll 25 participants. Participants will receive nilotinib BID and either 10, 15 or 20 mg of ruxolitinib BID. Maximum tolerated dose (MTD) of ruxolitinib will be determined.
  The second part of the trial will be a Phase II and will enroll 25 subjects. Participants will receive nilotinib and the MTD of ruxolitinib.
  Interventions: Drug: Nilotinib; Drug: Ruxolitinib

INTERVENTIONS:
Drug: Nilotinib — Nilotinib 300 mg BID
Drug: Ruxolitinib — Ruxolitinib, 10, 15 or 20mg BID

SUMMARY:
This study combines two drugs (ruxolitinib and the tyrosine kinase inhibitor, nilotinib) in an attempt to eliminate the CML (Chronic Myeloid Leukemia) stem cell population and thus allow for the deepest and most durable response possible in patients with CML in chronic phase who have achieved a complete hematologic remission (CHR), complete cytogenetic remission (CCyR), and major molecular remission (MMR), but not a complete molecular remission (CMR). The study will look at safety and tolerability of ruxolitinib when combined with nilotinib in a phase I study and will help establish the MTD (Maximum Tolerated Dose) of ruxolitinib when combined with nilotinib. Once the optimal dose of ruxolitinib is established in the phase I setting, a phase II evaluation will seek to establish the efficacy of this combination.

ELIGIBILITY:
Inclusion Criteria:

* Patients ≥ 18 years of age
* ECOG (Eastern Cooperative Oncology Group) Performance Status 0, 1, or 2
* Must have a diagnosis of Philadelphia chromosome positive (Ph+) chronic myeloid leukemia (CML) in chronic phase, with no previous evidence of accelerated or blast-phase disease.
* Must be actively receiving treatment for their CML with a tyrosine kinase inhibitor (TKI): imatinib, dasatinib, nilotinib or bosutinib, and must be on stable dose for > 1 year.
* Must have an ongoing complete hematologic response (CHR) on a TKI
* Must have an ongoing complete cytogenetic response (CCyR) on a TKI
* Must be in a major molecular remission (MMR) on a TKI for a minimum of 1 year leading up to enrollment.
* Adequate end organ function
* Adequate electrolytes
* Adequate platelet count
* Adequate neutrophil count
* Written informed consent prior to any screening procedures

Exclusion Criteria:

* Patients in complete molecular remission (CMR) on a TKI.
* Patients who have failed nilotinib or not tolerated nilotinib in the past
* Certain cardiovascular disorders
* Currently receiving treatment with strong CYP3A4 inhibitors which cannot be discontinued prior to starting study drug
* Actively receiving herbal medicines that are strong CYP3A4 inhibitors and/or inducers and treatment cannot be discontinued prior to starting study drug
* Currently receiving treatment with any medications that have the potential to prolong the QT interval that cannot be discontinued prior to starting study drug
* Impaired gastrointestinal (GI) function or GI disease that may significantly alter the absorption of the drug
* Acute or chronic pancreatic disease within the last year
* Cytopathologically confirmed Central Nervous System (CNS) infiltration
* Another primary malignancy that requires systemic chemotherapy or radiation
* Acute or chronic liver disease or severe renal disease considered unrelated to the cancer
* History of significant congenital or acquired bleeding disorder unrelated to cancer
* Major surgery within 4 weeks prior to Day 1 of the study or who have not recovered from prior surgery
* Past treatment with ruxolitinib
* Treatment with other investigational agent within 30 days of Day 1
* Inability to grant consent or history of non-compliance to medical regimens
* Women who are breastfeeding
* Women of child-bearing potential, unless they are using highly effective contraception

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2018-01 (Estimated); Primary Completion 2021-08 (Estimated); Study Completion 2021-08 (Estimated)

PRIMARY OUTCOMES:
Maximum Tolerated Dose (MTD) of ruxolitinib when combined with nilotinib | 2 Years
  Maximum Tolerated Dose (MTD) of ruxolitinib when combined with nilotinib
The number of patients that achieve a Complete Molecular Response (CMR) | 2 Years
  CMR is defined as an absence of the BCR-ABL1 transcript by qPCR performed on peripheral blood or bone marrow aspirate.

CONTACTS AND LOCATIONS:
Overall Officials: Patrick Burke, M.D., Principal Investigator — University of Michigan Rogel Cancer Center
Locations (2):
- United States (2):
  - The University of Michigan Comprehensive Cancer Center, Ann Arbor, Michigan
  - Wake Forest University Health Sciences, Winston-Salem, North Carolina